CLINICAL TRIAL: NCT06324838
Title: Extended Mesenteric Resection in Ileocecal Crohn's Disease to Prevent Recurrent Disease - A Randomized Controlled Trial.
Brief Title: Extended Mesenteric Resection in Ileocecal Crohn's Disease.
Acronym: EXCEED
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Odense University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 248-2021-NQ
Record Dates: First submitted 2023-08-21; First posted 2024-03-22 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Crohn's Disease of Terminal Ileum
Keywords: ileocecal resection; Mesocolic resection

STUDY DESIGN:
Intervention Model Description: Blinded multicenter randomized controlled clinical trial (RCT).
Who Masked: Participant, Care Provider
Masking Description: This randomized controlled trial will incorporate blinding procedures, with the understanding that due to the nature of this interventional surgical study, the operating surgeon cannot be blinded. However, rigorous measures will be implemented to ensure blinding of both patients and all other participants involved in patient treatment. The description of the surgery within the patient chart will follow a standardized format, with the exception of the resection details. Where the two treatment methods diverge, a predefined, standardized text referencing the study will be inserted.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Extended mesenteric resection (Experimental): Arm receiving ileocecal resection with extended mesenteric resection.
  Interventions: Procedure: Extended laparoscopic ileocecal resection
- Controls (Standard mesenteric resection) (Active Comparator): Arm receiving standard ileocecal resection.
  Interventions: Procedure: Standard laparoscopic ileocecal resection

INTERVENTIONS:
Procedure: Standard laparoscopic ileocecal resection — Participants will undergo standard mesocolic sparing resection.
  Other Names: Laparoscopic ileocecal resection
  Arms: Controls (Standard mesenteric resection)
Procedure: Extended laparoscopic ileocecal resection — Extended mesocolic resection to assess its impact on reducing recurrence at the anastomotic site.
  Arms: Extended mesenteric resection

SUMMARY:
The EXCEED project aims to study the role of the mesentery in disease recurrence in Crohn's disease (CD), as evidence suggests that including the mesentery when doing ileocecal resections can significantly reduce recurrence rates. The EXCEED study is a blinded randomised clinical trial with 204 participants having ileocecal Crohn's disease requiring resection. Participants will undergo either "standard" mesocolic sparing resection or extended mesocolic resection to assess its impact on reducing recurrence at the anastomotic site. The primary endpoint is endoscopic recurrence 12 months postoperatively.

Additionally, the study aims to evaluate the efficacy of different surveillance modalities in detecting anastomotic site recurrence. These examinations will be conducted pre- and postoperatively for a cohort of 20 participants.

Through this study, we seek to understand the mesentery's role in Crohn's disease recurrence and identify effective non-invasive methods for postoperative monitoring.

DETAILED DESCRIPTION:
Surgical Procedure and Perioperative Care Laparoscopic approach with a minimum 5 cm disease-free bowel on each side. Standard stapled side-to-side isoperistaltic anastomoses. Extended mesenteric excision involves resection of inflamed mesentery up to the level of visible inflammation.

Both treatment groups will receive standard postoperative care according to the standards of the hospital treating the participant.

Postoperative Follow-up Postoperative follow-up at 6 and 12 months. This consist of an ileo-colonoscopy, chart review and questionnaires. The early follow-up at 6 months aims to detect early recurrence, enabling early medical treatment or other intervention. The 12-month follow-up will be the primary endpoint to determine recurrence. Long-term outcomes will be assessed through a chart review after 3 and 5 years, documenting reoperations, clinical symptoms, pharmacological use, and other complications.

Postoperative Medicinal Use Postoperative medical prophylaxis assessment isn't explicitly detailed in the current protocol, though it will be acknowledged. Analysis will stratify participants based on pre- and post-operative biological/non-biological treatment. The treating physician will determine postoperative medical therapy, typically maintaining pre-operative medication.

Postoperative Endoscopy Endoscopy will be regarded as the golden standard for the detection of disease recurrence. The endoscopies, including bowel preparation and possible sedation, will be preformed in accordance with local guidelines at each hospital. At least three biopsies will be taken from the ileum (5 cm proximal to the anastomosis), anastomosis, and colon (5 cm below the anastomosis). A short video of each endoscopy will be saved for validation purposes. Lesions found during the endoscopy will be classified using the modified Rutgeerts score[7].

Patient-Reported Outcome During the preoperative workup (baseline), the participant will be asked to complete 2 questionnaires (5Q-5D-5L and SIBDQ). Postoperatively, the participant will be asked to complete the same questionnaires at 6 and 12 months.

Statistical analysis plan Outcome Analysis The investigators plan to conduct a chi-square or Fisher's exact test to compare the proportion of participants with endoscopic recurrence between the intervention and control groups.

The investigators will utilize logistic regression to adjust for potential confounding variables if needed.

Demographics The Investigators will use means and standard deviations (or medians and interquartile ranges) for continuous variables. For categorical variables, frequencies and percentages will be presented and demographic characteristics between intervention and control groups will be compared.

ELIGIBILITY:
Inclusion Criteria

* Patients above the age of 18 scheduled for ileocecal resection due to Crohn's disease.
* Relevant endoscopy and imaging within the last 6 months.
* Diagnosis of "simple" ileocecal Crohn's disease (limited to ileocecal disease with a maximum of 40 cm of affected ileum).

Exclusion Criteria

* Previous ileocecal resection.
* Inability to understand Danish or another Nordic language.
* Inability to comprehend the purpose and design of the project.
* Pregnancy or lactation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Estimated)
Dates: Start 2025-02-01 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2029-06 (Estimated)

PRIMARY OUTCOMES:
Endoscopic recurrence | 12 months postoperative
  Endoscopic signs of recurrence, defined as a modified Rutgeerts score >i2a.

SECONDARY OUTCOMES:
Early endoscopic recurrence | 6 months postoperative
  Endoscopic signs of recurrence, defined as a modified Rutgeerts score >i2a.
Clinical signs of recurrence / morbidity. | 6-48 months postoperatively
  Resumption of medicinal treatment. Chart review will be done to identify postoperative medicinal use.
Difference in disease severity | Perioperative
  At the time of operation according to the Montreal classification.
Patient reported outcome 1 | 6 and 12 months postoperative
  5Q-5D-5L
Patient reported outcome 2 | 6 and 12 months postoperative
  SIBDQ
Reoperations | 6 and 12 months postoperative
  Chart review will be done to identify any reoperations due to recurrence or other complications.
Perioperative complications | 30 days postoperative
  Postoperative complications according to Clavien-Dindo classification.
Cost of treatment | 12 months postoperative.
  Difference in treatment cost between the two groups. Reported in USD.

CONTACTS AND LOCATIONS:
Overall Officials: Mark B Ellebæk, PhD, Study Director — Surgical Research Unit, Odense University Hospital
Locations (1):
- Odense University Hospital, Odense, Denmark

IPD SHARING:
Plan to Share IPD: Yes
The principal investigators are committed to communicating the results, negative, positive, or inconclusive results, at local, national and international scientific meetings. The findings will be published in well-established, international peer-reviewed open access journals. After end of study, de-identified patient data will be uploaded to an open repository for further use.
Supporting Information: Study Protocol, SAP
Time Frame: After study completion.
Access Criteria: Available to all upon request

REFERENCES:
- [Derived] Baelum JK, Rosenberg J, Larsen P, Joergensen M, De La Croix H, Haglind E, Agenete E; BEAT-IBD research group; Kjeldsen J, Ellebaek MB. Extended mesenteric resection in Crohn's disease: EXCEED Study Protocol-a blinded multicenter randomized controlled clinical trial (RCT). Trials. 2025 Nov 21;26(1):532. doi: 10.1186/s13063-025-09261-3. PMID 41272703